CLINICAL TRIAL: NCT04753775
Title: RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED TRIAL OF ENEMA ALOE VERA GEL FOR ACHIVING REMISSION IN ACTIVE ULCERATIVE PROCTOSIGMOIDITIS.
Brief Title: RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED TRIAL OF ENEMA ALOE VERA GEL IN ACTIVE ULCERATIVE PROCTOSIGMOIDITIS.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Sandro Pertini, Roma (Other)
Responsible Party: Principal Investigator, Roberta Pica, MD, PhD, Ospedale Sandro Pertini, Roma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rif. 1836/11.03.10
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Aloe Vera Gel, Proctosigmoiditis, Remission, Trial, Ulcerative Colitis (UC)
MeSH Terms: conditions — Proctocolitis; Colitis, Ulcerative | interventions — Aloe vera gel

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: 22 patients were assigned to Group-A (5-ASA oral 800mg x 3 / day + 1 enema 60ml Aloe Vera gel / day) and 22 patients to Group-B (5-ASA oral 800mg x 3 / day + enema 60ml 1 Placebo / day).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 22 patients were assigned to Group-A (Experimental): 22 patients were assigned to Group-A
  Interventions: Drug: Aloe vera gel
- 22 patients were assigned to Group-B (Placebo Comparator): 22 patients were assigned to Group-B
  Interventions: Drug: Aloe vera gel

INTERVENTIONS:
Drug: Aloe vera gel

SUMMARY:
Aloe vera is used for the treatment of inflammatory bowel disease (IBD), but no data are present in regard the gel formulation as topical therapy in active ulcerative colitis.

DETAILED DESCRIPTION:
44 ulcerative colitis (UC) patients were enrolled and randomly allocated to treatment for 4 weeks with oral mesalazine (800 mg three times daily) and enema (60 ml aloe vera gel) 1/day (n = 22, Group A) or enema (60 ml placebo) (n = 22, Group B).

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years, mild to moderate active ulcerative proctosigmoiditis, diagnosed for the first time and no therapy started before. The maximum extension of the disease was accepted of 40-60 cm from the anal verge or distal disease.

Exclusion Criteria:

* an extension of disease above the sigma, renal impairment, pregnancy, lactation or established low compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-03-10 (Actual); Primary Completion 2010-04-10 (Actual); Study Completion 2010-05-10 (Actual)

PRIMARY OUTCOMES:
endoscopic remission | 4 weeks

IPD SHARING:
Plan to Share IPD: No